CLINICAL TRIAL: NCT05333471
Title: A Pilot Study of Fecal Microbiota Transplantation for Chronic Granulomatous Disease-Associated Colitis
Brief Title: Fecal Microbiota Transplantation for Chronic Granulomatous Disease-Associated Colitis
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10000809; 000809-I
Record Dates: First submitted 2022-04-15; First posted 2022-04-19 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01-26

CONDITIONS: Chronic Granulomatous Disease-associated Colitis
Keywords: Microbiome; Inflammation; Fecal Calprotectin; Immunodeficiency
MeSH Terms: conditions — Inflammation; Immunologic Deficiency Syndromes

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Interventional (Experimental): As this is a single arm study, this arm includes all participants. Participants will receive fecal microbiota transplantation (FMT) delivered by colonoscopy as a treatment for chronic granulomatous disease (CGD)-associated colitis (AC).
  Interventions: Drug: MTP 101-LF

INTERVENTIONS:
Drug: MTP 101-LF — Each unit of MTP-101-LF contains approximately 35 mL of fecal transplant product. Participants will receive approximately 32 mL via colonoscopy.

SUMMARY:
Background:

Chronic granulomatous disease (CGD) weakens the body's defense against germs. CGD can also damage the colon. It can cause inflammation (colitis) that disrupts the good bacteria. Placing good bacteria from donor stool into the intestine of a person with CGD (called fecal microbiota transplantation, or FMT) may help.

Objective:

To see if FMT can reduce inflammation in the colon.

Eligibility:

People aged 10-60 who have CGD and colitis, and the treatments they have tried are not helping or have side effects.

Design:

Participants will have a telehealth screening visit. They will have a medical record review and medical history. They will collect stool samples at home and mail them to NIH.

Participants will stay at the NIH hospital for 3-5 days. Each day, they will have the following:

Physical exam

Medical history and medicine review

Surveys about CGD and how it affects their life

Blood, stool, and urine tests

Participants will have a colonoscopy. They will be sedated. A long, flexible tube will be inserted into their rectum. The tube will deliver the FMT material to their colon. Small samples of intestinal tissue will be collected.

Participants may have an optional MRI of the digestive tract.

Participants will have 9 follow-up telehealth visits over 6 months. They will be asked about their symptoms and side effects. They will fill out short surveys. They will collect stool and urine samples at home. Up to 2 visits can be done in person. At these visits, they may have the option to have an MRI and another colonoscopy to get more tissue samples.

Participation will last for 6-7 months.

DETAILED DESCRIPTION:
Study Description:

This is a prospective, single-site, single-arm, open-label pilot trial to evaluate the use of fecal microbiota transplantation (FMT) delivered by colonoscopy as a treatment for chronic granulomatous disease (CGD)-associated colitis (AC). Participants will be evaluated for changes in intestinal inflammation, the microbiome, and symptoms associated with CGD-AC. It is hypothesized that FMT will reduce intestinal inflammation as measured by fecal calprotectin within 1 month compared to baseline (pre-FMT); there will be associated changes in the underlying stool microbiome and improvement in clinical symptoms.

Primary Objective:

To evaluate the change in intestinal inflammation pre-FMT vs post-FMT.

Secondary Objectives:

1. To evaluate the change in the stool microbiome pre-FMT vs post-FMT.
2. To evaluate changes in clinical symptoms pre-FMT and post-FMT.
3. Preliminary evaluation of the safety of FMT in CGD-AC.

Tertiary/Exploratory Objectives:

1. To evaluate other markers of intestinal and systemic inflammation pre-FMT and post-FMT.
2. To evaluate a washout period for beneficial effects of FMT on fecal calprotectin and the microbiome.
3. To evaluate the effect of FMT on antibiotic resistance in CGD-AC.

Primary Endpoint:

Difference in fecal calprotectin pre-FMT within 1 month post-FMT.

Secondary Endpoints:

1. Differences in alpha diversity, beta diversity, and relative abundance of taxa pre-FMT and within 1 month post-FMT. Assessment of engraftment of donor microbiome.
2. Difference in Patient Reported Outcome-2 (PRO-2) pre-FMT and within 1 month post-FMT.
3. Treatment-emergent adverse events (TEAEs).

Tertiary/Exploratory Endpoints:

1. Changes in C-reactive protein (CRP) and erythrocyte sedimentation rate (ESR) pre-FMT and post-FMT; changes in Simple Endoscopic Score for Crohn s Disease (SES-CD) pre-FMT and post-FMT in those who undergo a second colonoscopy; changes in magnetic resonance (MR) enterography findings in those who undergo a second MR enterography.
2. Changes in fecal calprotectin and microbiome indices over 6 months post-FMT.
3. Changes in antibiotic resistance genes in stool microbiome pre-FMT and post-FMT.

ELIGIBILITY:
* INCLUSION CRITERIA:

In order to be eligible to participate in this study, an individual must meet all of the following criteria:

1. Aged >=10 to <=60 years.
2. Able to provide informed consent (for ages >=18 years) or has a parent or guardian who can provide informed consent on their behalf (for ages <18 years).
3. Have confirmed prior diagnoses of CGD and CGD-AC (or CGD-IBD with evidence of colitis on colonoscopy).
4. Fecal calprotectin level >=200 microgram/g.
5. HBI score >=5 (to be evaluated on Day 1).
6. No planned change in systemic antibiotic regimen for CGD for 1 month preceding FMT.
7. No planned escalation in CGD-IBD treatment for 1 month preceding FMT.
8. If taking monoclonal antibodies for CGD-IBD, the dose must be stable for 12 weeks with no planned escalation.
9. Participants who can become pregnant must agree to use at least one highly effective method of contraception when engaging in sexual activities that can result in pregnancy, starting at screening until the end of study participation. Highly effective methods include a barrier (eg, condom, diaphragm, cervical cap), intrauterine device, or hormonal contraception.

EXCLUSION CRITERIA:

An individual who meets any of the following criteria will be excluded from participation in this study:

1. Evidence of acute GI infection, including active GI abscesses.
2. Presence of C difficile toxin gene in stool, as identified by PCR, in screening period.
3. History of intestinal obstruction definitively related to CGD-IBD.
4. History of fistulizing CGD-IBD or CGD-IBD intra-abdominal abscesses.
5. History of CGD-IBD related non-transversable intestinal strictures.
6. History of AEs attributable to previous FMT.
7. History of significant liver disease (eg, biopsy-proven nodular regenerative hyperplasia), including portal hypertension or cirrhosis.
8. Pregnant or breastfeeding.
9. History of severe food allergy.
10. Any contraindication to having colonoscopy under anesthesia.
11. Any condition that, in the opinion of the investigator, contraindicates participation in this study.

Ages: 10 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-08-08 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Difference in fecal calprotectin pre FMT and within 1 month post FMT. | Within 1 month
  To evaluate the change in intestinal inflammation pre-FMT vs post FMT

SECONDARY OUTCOMES:
Difference in PRO-2 pre-FMT and within 1 month post-FMT. | Within 1 month
  To evaluate the change in the stool microbiome pre-FMT vs post-FMT.
Differences in alpha diversity, beta diversity, and relative abundance of taxa pre-FMT within 1 month post-FMT and assessment of engraftment of donor microbiome and Assessment of engraftment of donor microbiome. | Within 1 month
  To evaluate the change in the stool microbiome pre-FMT vs post FMT.
Treatment-Emergent Adverse Events | Through end of study
  Preliminary evaluation of the safety of FMT in CGD-IBD.

CONTACTS AND LOCATIONS:
Overall Officials: Suchitra K Hourigan, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
Raw, de-identified data may be shared as part of publication. This may include microbiome and metabolome data.
Supporting Information: Study Protocol, ICF, CSR, Analytic Code
Time Frame: Exact time frame is unknown. Will be completed as part of publication requirements.
Access Criteria: Raw, de-identified data may be shared as part of publication. This may include microbiome and metabolome data. No other current plans for sharing exist.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_000809-I.html